CLINICAL TRIAL: NCT06339450
Title: Real World Environmental Exposure Study With Healthy and Cystic Fibrosis Subjects
Acronym: ExpoCF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ExpoCF
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis, Pulmonary
Keywords: cystic fibrosis; Environmental Exposure; exhaled breath condansate; Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase; level of hexanal; level of Neutrophil Elastase
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cystic fibrosis patients (Experimental): cystic fibrosis patient
  Interventions: Other: walk tours
- Patient Control (Experimental): patient without cystic fibrosis
  Interventions: Other: walk tours

INTERVENTIONS:
Other: walk tours — * During 5 days the patient will walk 4 hours in urban green space (open-space areas reserved for parks and other "green spaces", including plant life, water features -also referred to as blue spaces and other kinds of natural environment). The 3 hours walk tour includes a lunch break of one hour in the green space.
  * During 5 days the patient will walk 4 hours in urban space (including 3 hours walk around the city and one-hour lunch break.

SUMMARY:
Cystic fibrosis (CF) is the most common autosomal recessive disease that leads to early mortality in Caucasians and affects around 7500 patients in France. Progression of the disease depends on pulmonary exacerbations defined as acute deterioration of respiratory symptoms which ultimately impair lung function and quality of life. Most frequently caused by lung bacterial infections, exacerbations' effects include increased cough, increased sputum production, increased use of antibiotics, dyspnea and decreased lung function. The phenotypic variability of CF suggests the implication of other contributors especially to the CF airway disease. Beside genetic and epigenetic alterations, environmental factors - e.g tobacco smoke, air pollution, temperature changes, food intake - appear as relevant candidates. A previous review has discussed current knowledge on the effects of air pollution on the course of CF disease. Although scarce, the existing epidemiological andexperimental literature suggests a link between exposure to air pollutants and adverse health effects.Although scarce, the existing epidemiological and experimental literature suggests a link between exposure to air pollutants and adverse health effects. The EU sponsored REMEDIA project (Impact of exposome on the course of lung diseases, Grant agreement ID 874753) contributes to the understanding of the influence of the exposome on chronic obstructive pulmonary disease (COPD) and CF. Objective of work package 3 within the REMEDIA project is the development of a mobile environmental sensor toolbox that is capable to assess the external exposome. The biomarkertoolbox was developed and tested in a proof-of-concept study carried out in healthy volunteers. The next step is to validate the collectionof exhaled breath condensate (EBC) in a real-life study. In this aim, the objective of the present study will be to assess the feasibility of EBC collection in CF patients and healthy individuals

ELIGIBILITY:
Inclusion Criteria:

* Normal blood test
* Negative Cotinine test
* Protocole (RiPH2)
* Normal ECG
* Normal alcohol test
* Lung function with FEV1 predicted ≥ 40% at spirometry.

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Collection of exhaled breath condensate (EBC) for biomarker analysis | day 1
  Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase in EBC
Collection of exhaled breath condensate (EBC) for biomarker analysis | days 3
  Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase in EBC
Collection of exhaled breath condensate (EBC) for biomarker analysis | days 5
  Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase in EBC
Collection of exhaled breath condensate (EBC) for biomarker analysis | days 6
  Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase in EBC
Collection of exhaled breath condensate (EBC) for biomarker analysis | days 8
  Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase in EBC
Collection of exhaled breath condensate (EBC) for biomarker analysis | days 10
  Levels of 3-Nitrotyrosin, Hexanal, Neutrophil Elastase in EBC

SECONDARY OUTCOMES:
Dysfunction or misused, failure, of EBC and sensor device | days 10
  rate of Dysfunction or misused, failure, of EBC and sensor device
Show correlation of biomarker signal with environmental sensor system in a clinical challenge setting in healthy and CF patients. | days 5
  Correlation of environmental exposome signal biomark
Describe differences in CF subjects vs. healthy controls | days 5
  Comparison of environmental exposome signal biomarker and environmental sensor measures in healthy individuals and CF patients
Impact of environment exposome on health status and lung function | days 5
  Lung function testing and health questionnaire score before and after working trial in urban and green zone
Show correlation of biomarker signal with environmental sensor system in a clinical challenge setting in healthy and CF patients. | days 10
  Correlation of environmental exposome signal biomark
Describe differences in CF subjects vs. healthy controls | days 10
  Comparison of environmental exposome signal biomarker and environmental sensor measures in healthy individuals and CF patients

CONTACTS AND LOCATIONS:
Overall Officials: ralph Epaud, Principal Investigator — CHI CRETEIL